CLINICAL TRIAL: NCT00778310
Title: Functional Neuroimaging of Acute Concerta Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD): Differences Across Development
Brief Title: Neuroimaging of the Effects of Concerta in the Treatment of ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CONCERTAATT4087
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concerta (Experimental): The subject will be administered their usual dose of Concerta the morning of the FMRI scan in a double blind fashion
  Interventions: Drug: methylphenidate-OROS
- Placebo (Placebo Comparator): The subject will be administered a placebo the morning of the FMRI scan in a double blind fashion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate-OROS — The collaborator (Ortho-McNiel Janssen Scientific Affairs, LLC) will provide capsules of Concerta that are made to appear similar to placebo capsules. The subject will be administered their usual dose of Concerta the morning of the scan.
  Arms: Concerta
Drug: Placebo — The collaborator (Ortho-McNiel Janssen Scientific Affairs, LLC) will provide capsules of placebo that are made to appear similar to Concerta capsules. The subject will be administered placebo the morning of the scan.
  Arms: Placebo

SUMMARY:
A number of brain regions have been down to be altered in both structure and function in patients with ADHD, including prefrontal cortex, anterior cingulate, caudate and cerebellum. Patients with ADHD often show reduced levels of activity in the frontal and cingulate regions of brain while performing measures of inhibitory control during functional magnetic resonance imaging (fMRI). While stimulant medications robustly improve the clinical symptoms of ADHD, there are only a small number of studies examining the effects of these commonly prescribed medications on brain activity. We propose to obtain fMRI in patients with ADHD on placebo and on their individualized dose of OROS methylphenidate (Concerta). Our hypothesis is that Concerta will increase the activity of the brain in the frontal, cingulate and amygdala of the brain and that these brain changes will be associated with clinical improvement of symptoms.

DETAILED DESCRIPTION:
Three age groups of subjects will be studied: school age children (aged 9-12), older adolescents (age 15-17 years) and young adults (age 20-25 years). Twenty subjects will be studied in each group. All subjects must meet criteria for ADHD, combined type and be either treatment naïve or currently taking and responding well to Concerta. Child and adolescent patients taking Concerta will have their current levels of ADHD symptoms assessed with the Dupaul ADHD rating scale (11); adults taking Concerta will be assessed with Conners Adult ADHD Rating Scale (CAARS). Patients whose symptoms are in remission as evidenced by scores in the normal range on these scales may proceed directly to the neuroimaging portion of the study. Subjects who are treatment naïve or are treated but are not in remission shall under a three week open label trial of Concerta to determine the optimal dose for treatment of their symptoms.

Subjects will have two fMRI sessions on different days. During each fMRI session, they will perform both the Stop Signal Task and the Emotional Conflict Resolution Task . On the morning of the scan, placebo and Concerta will be administered in a double-blind, crossover design, with order of medication and placebo randomized. The scan sessions will take place between 3 and 7 hours after medication administration. After each scan, the subject and a research assistant will go to a quiet room in the imaging center; the subjects will be given arithmetic level set at a level of difficulty that the subject has mastered. The subject will be given 15 minutes to complete as many problems as possible.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Attention Deficit Hyperactivity Disorder
* Current clinical responder to Concerta (OROS-methylphenidate)

Exclusion Criteria:

* IQ < 95
* Presence of Learning Disorder
* Presence of an Affective or Psychotic Disorder
* Presence of a Substance/Alcohol Abuse/Dependence Disorder
* Presence of an Autism Spectrum Disorder
* Presence of a Tic Disorder
* Taking any psychotropic medication other than Concerta
* A medical condition requiring daily medication
* Previous adverse or non response to Concerta

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Pliszka, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Dept of Psychiatry, UTHSCSA, San Antonio, Texas, United States

REFERENCES:
- [Background] Bush G, Spencer TJ, Holmes J, Shin LM, Valera EM, Seidman LJ, Makris N, Surman C, Aleardi M, Mick E, Biederman J. Functional magnetic resonance imaging of methylphenidate and placebo in attention-deficit/hyperactivity disorder during the multi-source interference task. Arch Gen Psychiatry. 2008 Jan;65(1):102-14. doi: 10.1001/archgenpsychiatry.2007.16. PMID 18180434
- [Background] Pliszka SR, Glahn DC, Semrud-Clikeman M, Franklin C, Perez R 3rd, Xiong J, Liotti M. Neuroimaging of inhibitory control areas in children with attention deficit hyperactivity disorder who were treatment naive or in long-term treatment. Am J Psychiatry. 2006 Jun;163(6):1052-60. doi: 10.1176/ajp.2006.163.6.1052. PMID 16741206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 75 patients were enrolled from 11/4/2008 t0 8/12/2010. Patients were recruited from advertisements in local papers as well as flyers in the UTHSCSA psychiatric clinic.
Pre-assignment Details: Psychiatric assessment was performed to confirm the diagnosis of ADHD. Fifteen (15) patients were screen failures. Five (5) patients did not respond to an open label trial of Concerta were excluded. 11 withdrew consent or lost to follow up. (1) withdrew to claustrophobia. 43 were exposed to study drug (Concerta and placebo) in crossover design.
Groups:
- Adults: These were participants between the age of 21-25 years. They underwent 2 FMRI studies, once on placebo and once on Concerta in a double blind randomized crossover design.
- Children: These were participants between the age of 3- 17 years. They underwent 2 FMRI studies, once on placebo and once on Concerta in a double blind randomized crossover design.
Period: Overall Study
Arm/Group | Adults | Children
Started | 17 | 26
Usable Data | 14 | 21
Completed | 17 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults | Children | Total
Number analyzed (Participants) | 17 | 26 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 26 | 26
  Between 18 and 65 years | 17 | 0 | 17
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.2 (1.78) | 11.3 (2.1) | 15.6 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  United States | 17 | 26 | 43

OUTCOME MEASURES:

1. Primary Outcome: Brain Oxygenation Level Dependent Signal in the Fusiform Gyrus and the Amygdala on Concerta vs. Placebo
Description: Each subject viewed shapes and faces on multiple trials. The subject matched faces or shapes on each trial. BOLD activity during shape trials was subtracted from BOLD activity during Face trials and this value was compared on drug vs. placebo trials.
Time Frame: Placebo and Drug day, 1-2 weeks apart
Population: The number who completed both fMRI one week apart (crossover study, scanned twice
Measure: Mean (Standard Deviation); unit: Face-Shape BOLD signal difference
Groups:
- Adults Drug Condition; Children Drug Condition: This is the BOLD signal data on the Concerta day scan.
- Adults Placebo Condition; Children Placebo Condition: This is the BOLD signal data on the Placebo day scan.
Arm/Group | Adults Drug Condition | Adults Placebo Condition | Children Drug Condition | Children Placebo Condition
Number analyzed (Participants) | 14 | 14 | 21 | 21
Face-Shape BOLD signal difference
  Amygdala | 1.79 (1.06) | 0.58 (1.09) | 1.43 (1.08) | 0.77 (1.36)
  Fusiform Gyrus | 1.46 (1.36) | 1.64 (1.21) | 1.99 (1.1) | 1.06 (1.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on the day of the scans.
Arm/Group | Adults | Children
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/26
Other Adverse Events (participants affected / at risk) | 0/17 | 0/26

LIMITATIONS AND CAVEATS:
No typically developing control group compared to either the adult or child group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No